CLINICAL TRIAL: NCT03611192
Title: Effects of A Multicomponent Exercise on Executive Function and Balance in Pre-frail Older Adults
Brief Title: Multicomponent Exercise on Executive Function and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM107051F
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Health Services for the Aged
Keywords: Multicomponent Exercise; Executive Function; Balance; Pre-frail

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise group (Experimental)
  Interventions: Other: Multicomponent exercise
- Home-program exercise group (Active Comparator)
  Interventions: Other: Home-program exercise

INTERVENTIONS:
Other: Multicomponent exercise — Aerobic exercise: 15~20 mins Resistance exercise: 15 mins Balance exercise: 15~20 mins Flexibility exercise: 10 mins
  Arms: Multicomponent exercise group
Other: Home-program exercise — 60 mins exercise
  Arms: Home-program exercise group

SUMMARY:
The present study is to examine the effects of a multicomponent exercise on executive function and balance in pre-frail older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 65
* Pre-frail according to the Fried Physical Frailty Phenotype
* Community-dwelling and able to walk independently>6m

Exclusion Criteria:

* Unstable medical condition (ACSM Health Facility Pre-participation Screening Questionnaire)
* Neurological conditions(eg, Parkinson's disease, stroke, multiple sclerosis)
* MMSE<24
* Visual or color discrimination impairment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Trail-Making test | Change from baseline at 12 weeks
  Executive function
Stroop test | Change from baseline at 12 weeks
  Executive function
Digit span test | Change from baseline at 12 weeks
  Executive function
Mini-Balance Evaluation Systems Test | Change from baseline at 12 weeks
  Balance
Time Up & Go test | Change from baseline at 12 weeks
  Balance
One leg standing test | Change from baseline at 12 weeks
  Balance

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Change from Baseline at 12 weeks
  Global cognition
Fried frailty criteria | Change from baseline at 12 weeks
  Frailty reverse

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan